CLINICAL TRIAL: NCT04339582
Title: GENETIC BASIS of LEFT VENTRICULAR APICAL HYPOPLASIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Monaldi Hospital (Other)
Collaborators: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, GIUSEPPE LIMONGELLI, Principal Investigator, Monaldi Hospital
Other Study IDs: LVAH_001
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Left Ventricular Apical Hypoplasia (LVAH), New Rare Condition
Keywords: Left ventricular apical hypoplasia (LVAH); Genetic testing; Congenital or genetical condition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brief summary Left ventricular apical hypoplasia (LVAH) is a rare cardiomyopathy characterized by a spherical, truncated LV with some degree of systolic dysfunction, an elongated, normally functioning right ventricle that wraps around the distal left ventricle, deficiency of the myocardium within the LV apex with adipose tissue infiltrating the apex and origin of the papillary muscle in the flattened anterior apex. This condition presents with different clinical presentation, ranging from no symptoms to congestive heart failure or malignant tachycardia. The etiology of this condition is currently unknown. The aim of this study is to evaluate the clinical and genetic characteristics of patients with LVAH.

Background Left ventricular apical hypoplasia (LVAH) is described as congenital heart disease with an unusual type of cardiomyopathy that was first described in 2004 by Fernandez-Valls et al. It is an extremely rare disease; to date, only more than twenty cases were described.

The typical imaging features of this cardiomyopathy include: a spherical, truncated LV with some degree of systolic dysfunction; an elongated, normally functioning right ventricle that wraps around the distal left ventricle; deficiency of the myocardium within the LV apex with adipose tissue infiltrating the apex; origin of the papillary muscle in the flattened anterior apex. A 2D echocardiogram and cardiac MRI can successfully indicate different morphological features This rare phenomenon frequently presents with different clinical manifestations according to the age of the disease, from no symptoms in children to congestive heart failure, pulmonary edema, or even malignant tachycardia in adults. Congenital or genetical etiology was proposed to explain the development of this rare cardiomyopathy.

The aim of this study is to evaluate the clinical and genetic characteristics of patients with LVAH.

Methods Study population

The study population is composed by consecutive patients with diagnosis of LVAH. Diagnosis of LVAH is based on echocardiographic or cardiac magnetic resonance (CMR) evidence of all the following diagnostic criteria:

* a spherical, truncated LV with some degree of systolic dysfunction;
* an elongated, normally functioning right ventricle that wraps around the distal left ventricle;
* deficiency of the myocardium within the LV apex with adipose tissue infiltrating the apex;
* origin of the papillary muscle in the flattened anterior apex. Patients enrolled followed a common protocol designed by GL (Monaldi Hospital, AORN Colli, University of Campania "Luigi Vanvitelli"). The study protocol was approved, and written informed consent was obtained from each subject, according to the procedure established by the Ethic Committee of our institution.

Study protocol Patients enrolled underwent a comprehensive clinical-genetic evaluation commonly practiced in our cardiology division. In particular, the basal evaluation, consisted family and personal history, physical examination, blood tests, 12-lead electrocardiogram (ECG) at rest, conventional M-mode, two-dimensional and Doppler echocardiography, 24-hour Holter ECG, and cardiac magnetic resonance (CMR), and genetic testing with whole exome sequencing (WES). Moreover, all patients are clinically revaluated every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 0-90 years old, in any distribution.
* Patients who have the diagnostic criteria for LVAH. Diagnosis of LVAH is based on echocardiographic or cardiac magnetic resonance (CMR) evidence of all the following diagnostic criteria:

  * a spherical, truncated LV with some degree of systolic dysfunction;
  * an elongated, normally functioning right ventricle that wraps around the distal left ventricle;
  * deficiency of the myocardium within the LV apex with adipose tissue infiltrating the apex;
  * origin of the papillary muscle in the flattened anterior apex.

Exclusion Criteria:

* Involvement with any other ongoing studies.
* Patients who have diagnosis of other Cardiomyopathies

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed by consecutive patients with diagnosis of LVAH. Diagnosis of LVAH is based on echocardiographic or cardiac magnetic resonance (CMR) evidence of all the following diagnostic criteria:
  * a spherical, truncated LV with some degree of systolic dysfunction;
  * an elongated, normally functioning right ventricle that wraps around the distal left ventricle;
  * deficiency of the myocardium within the LV apex with adipose tissue infiltrating the apex;
  * origin of the papillary muscle in the flattened anterior apex. Patients enrolled followed a common protocol designed by GL (Monaldi Hospital, AORN Colli, University of Campania "Luigi Vanvitelli"). The study protocol was approved, and written informed consent was obtained from each subject, according to the procedure established by the Ethic Committee of our institution.
Sampling Method: Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2013-09-20; Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
new gene of LVAH | one year later the completation study
  the principal aim of the study is to identify the new gene of LVAH and to investigate on genetic background of this clinical condition

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale V. Monaldi, Università degli studi della Campania, Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No